CLINICAL TRIAL: NCT06190587
Title: The Evaluation of the Impact of Goji Berry Consumption Some Biochemical Parameters in Healthy Individuals
Brief Title: Effect of Goji Berry Consumption on Biochemical Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-22/01
Record Dates: First submitted 2023-11-01; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Hyperlipidemias
Keywords: Functional Food; Goji Berry; Serum Lipids; Serum Fasting Glucose
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): In control group participants had 8-weeks follow-up without any intervention.
- Interventional Group (Experimental): In interventional group participants had 8-weeks follow-up with 20 g/day goji berry consumption intervention.
  Interventions: Dietary Supplement: Goji Berry

INTERVENTIONS:
Dietary Supplement: Goji Berry — As a functional food goji berry contains 19 amino acids, 21 minerals, a wide range of carotenoids (β-Carotene, Neoxanthin, Cryptoxanthin, Zeaxanthin), polysaccharides, flavonoids, phytosterols, vitamin A, C and E.
  Arms: Interventional Group

SUMMARY:
Goji Berry as a functional food have been shown to reduce risk of hyperlipidemia, type 2 diabetes, etc. However, human studies are limited in this area. In this study, it has been aimed to evaluate the effect of goji berry consumption on some biochemical parameters in healthy individuals.

DETAILED DESCRIPTION:
Healthy individuals have been divided into control and study groups. Individuals in both group have same characteristics such as age, gender, and body mass index (Control Group: 35 individuals - Study Group: 35 individuals). Both group were asked to maintain their normal diets. In addition, the study group consume 20 g of dried goji berry per day and did not consume any fruit with a similar antioxidant content during the 8 weeks study period. The control group was asked to exclude goji berry and similar fruits with high antioxidant content from their diet during the 8 weeks study period. The 20 g goji berry for per day was given weekly to each individual in a study group in transparent bags. At the beginning of the study and every 15 days, food consumption record for 3 consecutive days (2 weekdays and 1 weekend), a 3-day physical activity record, and anthropometric measurements (weight, height, waist and hip circumferences, body composition analysis) were taken. Blood parameters (total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL), very low density lipoprotein (VLDL), triglyceride, glucose, insulin, homeostatic model assessment of insulin resistance (HOMA-IR), HbA1c) of individuals were taken at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20-25 kg/m²
* Female individuals are not in the period of lactation and menopause,
* Absence of any chronic or acute disease diagnosed by a physician,
* No allergies to Goji Berry
* Not consuming goji berry and similar fruits regularly for the last 1 month.
* Not being in the process of body weight loss
* Not doing strenuous physical activity
* Not taking any medication or antioxidant vitamin support
* Not smoking
* Not consuming alcohol (moderate alcohol consumption)

Exclusion Criteria:

Not meeting the criteria for inclusion in the study

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
serum lipids | 8 weeks
  change in serum lipids level in interventional group.
fasting glucose | 8 weeks
  change in fasting glucose levels in interventional group.
serum insulin | 8 weeks
  change in serum insulin levels in interventional group.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Turkish Republic of Northern Cyprus, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided